CLINICAL TRIAL: NCT01878539
Title: Oral Anticoagulation and Self-management: Analysis of the Factors That Determine the Feasibility of Using Self-testing and Self-management in Primary Care
Brief Title: Oral Anticoagulation and Self-management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osakidetza (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Eduardo Tamayo Aguirre, Family Doctor, Osakidetza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ISCIII-11/02285
Record Dates: First submitted 2013-06-07; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Atrial Fibrillation; Embolism
MeSH Terms: conditions — Atrial Fibrillation; Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health Center training (Experimental): The intervention will consist of a patient training programme involving the provision of information and practical training concerning their condition and its treatment, as well as how to use a portable blood coagulation monitoring device and adjust their anticoagulant dose.
  Interventions: Device: coagulometer; Behavioral: training programme

INTERVENTIONS:
Device: coagulometer
  Other Names: how to use a portable blood coagulation monitoring device and adjust their anticoagulant dose
Behavioral: training programme
  Other Names: patient training programme involving the provision of information and practical training concerning their condition and its treatment

SUMMARY:
An intervention program targeting patients and caregivers based on education about their condition and training in the use of portable coagulomenter to self monitor and training on the treatment adjustment to self manage, can be effective to enable patients in OACs to self manage as well as to identify determinant factors associated with the success and failure of the program.

DETAILED DESCRIPTION:
BACKGROUND: The skills of patients on oral anticoagulants are critical for achieving good outcomes with this treatment. Self-management, or the capacity of patients to control their INR (International Normalized Ratio)level and adjust their treatment, is an effective strategy of treatment. Capacity of patients to self manage is determined by a range of factors. The identification of these factors would improve the design of self management programmes and in turn increase the number of patients able to self-manage. The objective of our study is to identify those factors that determine the ability of patients on oral anticoagulant therapy to achieve self-management of their treatment.

METHOD: This will be a three year quasi- experimental prospective study with a control group. 333 patients on anticoagulant therapy from five health centres of the Basque Health Service are to be followed up for a period of six months each after the intervention, to assess their ability to self-test and self-manage. The intervention will consist of a patient training programme involving the provision of information and practical training concerning their condition and its treatment, as well as how to use a portable blood coagulation monitoring device and adjust their anticoagulant dose.

DISCUSSION: Training programmes for self-management are effective in terms of enabling patients to acquire the necessary skills, though the level of success seems to depend on various patient-related factors. Given the proven benefits of self-management, it would be useful to properly characterise these factors and use this information to successfully increase the percentage of patients on on oral anticoagulants able to self-manage their own treatment.

ELIGIBILITY:
Inclusion Criteria:

* Anticuagulated
* Living in the study area

Exclusion Criteria:

* Older than 16 years old
* More than one year cuagulated

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Control of INR (International Normalized Ratio) | 6 months
  So the primary objectives of this study are to assess the ability of patients/caregivers to test INR (International Normalized Ratio) levels with a portable coagulometer and capillary whole blood from a finger prick and the impact of a range of factors on the ability of patients on OACs to self-monitor and self-manage their treatment.
  If the INR is within the personal range above 80% it will consider a good control

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tamayo, Doctor, Principal Investigator — Osakidetza
Locations (1):
- Osakidetza, Donostia / San Sebastian, Gipuzkoa, Spain

REFERENCES:
- [Derived] Tamayo Aguirre E, Galo-Anza A, Dorronsoro-Barandiaran O, Del Burgo EU, Ostiza Irigoyen A, Garcia-Carro A, Lopez-Fernandez I, Colera N, Saez-Garbayo P, Tamayo-Uria I. Oral anticoagulation with vitamin K inhibitors and determinants of successful self-management in primary care. BMC Cardiovasc Disord. 2016 Sep 13;16(1):180. doi: 10.1186/s12872-016-0326-z. PMID 27624485
- [Derived] Tamayo Aguirre E, Vergara-Mitxeltorena I, Uranga Saez Del Burgo E, Ostiza-Irigoyen A, Garcia-Carro A, Lopez-Fernandez I, Galo-Anza A. Oral anticoagulation and self-management: analysis of the factors that determine the feasibility of using self-testing and self-management in primary care. BMC Cardiovasc Disord. 2013 Aug 22;13:59. doi: 10.1186/1471-2261-13-59. PMID 23968316